CLINICAL TRIAL: NCT02022631
Title: Comparison Between Standard and New Alternative Formats of the Summary-of-Findings Tables in Cochrane Review Users. A Non-inferiority Randomized Controlled Trial
Brief Title: New Alternative Formats vs Standard of SoF Tables. Non-inferiority Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Holger Schunemann, MD, MSc, PhD, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MIF_aim1RCT1
Record Dates: First submitted 2013-12-13; First posted 2013-12-30 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: GRADE Approach; Summary of Findings Table; Cochrane Collaboration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alternative SoF (Experimental): Investigators will compare one SoF table with alternative formats (Table A) against one SoF table with the current formats (Table B). In both tables, the clinical question in terms of patients and setting, intervention, comparator, and outcomes informed by the tables, and the complementary information included as footnotes will be the same. The only differences between the current and alternative SoF table formats will be different methods to either show the same data in a different way or to provide complementary data to the one showed in the current format (i.e. supplementary data as risk difference).
  Interventions: Other: Alternative summary of findings table format
- Current SoF (Active Comparator): Investigators will compare one SoF table with alternative formats (Table A) against one SoF table with the current formats (Table B). In both tables, the clinical question in terms of patients and setting, intervention, comparator, and outcomes informed by the tables, and the complementary information included as footnotes will be the same. The only differences between the current and alternative SoF table formats will be different methods to either show the same data in a different way or to provide complementary data to the one showed in the current format (i.e. supplementary data as risk difference).
  Interventions: Other: Current summary of findings table format

INTERVENTIONS:
Other: Alternative summary of findings table format — Investigators will compare one SoF table with alternative formats (Table A) against one SoF table with the current formats (Table B). In both tables, the clinical question in terms of patients and setting, intervention, comparator, and outcomes informed by the tables, and the complementary information included as footnotes will be the same. The only differences between the current and alternative SoF table formats will be different methods to either show the same data in a different way or to provide complementary data to the one showed in the current format (i.e. supplementary data as risk difference).
  Arms: Alternative SoF
Other: Current summary of findings table format — Investigators will compare one SoF table with alternative formats (Table A) against one SoF table with the current formats (Table B). In both tables, the clinical question in terms of patients and setting, intervention, comparator, and outcomes informed by the tables, and the complementary information included as footnotes will be the same. The only differences between the current and alternative SoF table formats will be different methods to either show the same data in a different way or to provide complementary data to the one showed in the current format (i.e. supplementary data as risk difference).
  Arms: Current SoF

SUMMARY:
The investigators will conduct a parallel two-armed, non-inferiority randomized trial comparing new alternative formats of summary of findings tables (SoF) tables with current formats. The investigators will contact Cochrane review users by email and will ask them to fill a questionnaire developed using the "Survey Monkey" online system. The survey will include questions about baseline information (demographic characteristics, background, number of visits to the Cochrane Library, familiarity with the GRADE system, etc.). Then, participants will be stratified (health professional, guideline developer, researcher) and randomly assigned to one of the two SoF table formats, either the alternative (Table A) or the current one (Table C). Participants will be asked to answer questions to determine understanding, accessibility, and satisfaction with the formats to which they were randomized. Finally, the investigators will show them the table format to which they were not initially allocated in order to test their preference for either one.

ELIGIBILITY:
Inclusion Criteria:

* Cochrane review users
* Authors of systematic reviews
* Health professionals
* Guideline developers
* Researchers

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Understanding of key findings | 30 minutes
  Investigators will frame multiple-choice questions about key concepts in the table with five response alternatives for each question and only one correct answer. Then, investigators will compare the proportion of correct answers between groups per question

SECONDARY OUTCOMES:
Accessibility of information | 30 minutes
  This outcome will consider 3 domains: (1) how easy is to find critical information in the table, (2) how easy is to understand the information, and (3) whether the information is presented in a way that is helpful for decision-making. These three domains will be measured presenting to participants three statements to which they have to indicate the degree of agreement: "It was easy to find the information about the effects", "It was easy to understand the information", and "The information is presented in a way that would help me make a decision" using a 7-point Likert scale (1= I strongly disagree, 2= I disagree, 3= I somewhat disagree, 4= Not sure, 5= I somewhat agree, 6= I agree, and 7= I strongly agree). The outcome overall accessibility of information will be obtained as the average of responses for each domain, per participant.
Overall satisfaction | 30 minutes
  It will be measured using a 7-point Likert scale with 3 anchors: 1= strongly dissatisfied, 4= neither satisfied nor dissatisfied, 7= strongly satisfied, and it will be treated as a continuous outcome. Investigators will compare the means per group.
Preference | 30 minutes
  This outcome taps the question: Between alternative (Table A) and current format (Table B) of SoF table, "which table does the user prefer?" It will be measured using a 5-point Likert scale (1= strongly prefer table B, 2= I prefer table B, 3= Both table A and B are good to me, 4= I prefer table A, 5= I strongly prefer table A), and it will be treated as continuous outcome. Investigators will describe the data obtained in each group. Other questions related to participants' preference for each alternative item will be included.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Schünemann, MD, MSc, PhD, Principal Investigator — McMaster University; Alonso Carrasco-Labra, DDS, MSc, Study Director — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrasco-Labra A, Brignardello-Petersen R, Santesso N, Neumann I, Mustafa RA, Mbuagbaw L, Etxeandia Ikobaltzeta I, De Stio C, McCullagh LJ, Alonso-Coello P, Meerpohl JJ, Vandvik PO, Brozek JL, Akl EA, Bossuyt P, Churchill R, Glenton C, Rosenbaum S, Tugwell P, Welch V, Garner P, Guyatt G, Schunemann HJ. Improving GRADE evidence tables part 1: a randomized trial shows improved understanding of content in summary of findings tables with a new format. J Clin Epidemiol. 2016 Jun;74:7-18. doi: 10.1016/j.jclinepi.2015.12.007. Epub 2016 Jan 11. PMID 26791430
- [Derived] Carrasco-Labra A, Brignardello-Petersen R, Santesso N, Neumann I, Mustafa RA, Mbuagbaw L, Ikobaltzeta IE, De Stio C, McCullagh LJ, Alonso-Coello P, Meerpohl JJ, Vandvik PO, Brozek JL, Akl EA, Bossuyt P, Churchill R, Glenton C, Rosenbaum S, Tugwell P, Welch V, Guyatt G, Schunemann H. Comparison between the standard and a new alternative format of the Summary-of-Findings tables in Cochrane review users: study protocol for a randomized controlled trial. Trials. 2015 Apr 16;16:164. doi: 10.1186/s13063-015-0649-6. PMID 25873338
- See also: Related Info — http://www.cochrane.org
- See also: Related Info — http://www.gradeworkinggroup.org